CLINICAL TRIAL: NCT07064083
Title: The Effect of Intra-Canal Ketorolac Application on Post-Endodontic Pain: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Intra-Canal Ketorolac Application on Post-Endodontic Pain
Acronym: Post-Endodonti
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sabah Morad Sobhy, Endodontic department, al azhar university, cairo, Egypt., Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/0036
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: To Evaluate the Effectiveness of Intra-canal Nano-ketrolac as a Medicament in Reducing Post-endodontic Pain in Patients Undergoing Root Canal Treatment
Keywords: postendodontic pain; nano-ketrolac

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo-controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GI (Experimental): The nano-ketrolac gel will be introduced intracanal after cleaning and shaping is performed.
  Interventions: Drug: intracanal nano-ketrolac
- GII (Experimental): ketrolac gel will be introduced intracanal after cleaning and shaping is performed.
  Interventions: Drug: ketrolac gel
- GIII (Placebo Comparator): A placebo gel will be introduced intracanal after cleaning and shaping is performed.
  Interventions: Drug: A placebo gel

INTERVENTIONS:
Drug: intracanal nano-ketrolac — For the subjects of GI nano-ketorolac gel (Around 2mm3), placed as medicament inside the root canal for one week. The obturation through cold lateral compaction technique is to be carried out on the next visit.
  Arms: GI
Drug: ketrolac gel — For the subjects of GII, ketorolac gel (Around 2mm3), placed as medicament inside the root canal for one week. The obturation through cold lateral compaction technique is to be carried out on the next visit.
  Arms: GII
Drug: A placebo gel — a placebo gel is placed and retained for one week. The obturation through cold lateral compaction technique is to be carried out on the next visit.
  Arms: GIII

SUMMARY:
After obtaining informed consent, the procedure begins with the administration of local anesthesia to ensure patient comfort. A standard approach involves using 2% lidocaine with 1:100,000 epinephrine, delivered either via infiltration for maxillary teeth or mental nerve block for mandibular posterior teeth. Adequate anesthesia is confirmed using a cold test or gentle probing. Once profound anesthesia is achieved, rubber dam isolation is placed to maintain an aseptic field and prevent contamination. The operative field is then disinfected with 5% sodium hypochlorite before proceeding to the access cavity preparation.

The access cavity is prepared using a high-speed diamond bur under continuous water coolant. The shape of the access cavity is determined by the tooth's anatomy, ensuring straight-line access to the canal system. Once the pulp chamber is opened, the roof is carefully removed using a round bur or ultrasonic tips, exposing the canal orifices. The chamber is then thoroughly irrigated with 2.5% sodium hypochlorite to remove any residual pulp tissue and debris. A DG16 endodontic explorer is used to locate the canal orifices, after which initial canal exploration is performed using a #10 or #15 K-file to check for patency.

Working length determination follows, utilizing an electronic apex locator (EAL) to establish the length of the canal. A confirmation periapical radiograph is taken to verify the readings. To maintain apical patience, a #10 K-file is used in a gentle watch-winding motion until it reaches the apical constriction. The glide path is then established to facilitate subsequent instrumentation. This is achieved by sequentially using hand files (#10, 15, and 20 K-files) with a balanced force technique until a #20 file moves freely to the working length. Throughout this process, frequent irrigation with 2.5% sodium hypochlorite is performed to flush out debris and maintain canal cleanliness.

Once the glide path is established, shaping of the canal begins based on the size of the initial binding file, which is the first file to engage the canal walls at the working length. If the initial binding file is #10 or #15, the apical preparation is typically completed up to a size #35, while an initial binding file of #20 may require enlargement to #40 or #50. Canal shaping is performed using a crown-down technique with rotary nickel-titanium (NiTi) instruments.

Throughout the shaping process, continuous irrigation with sodium hypochlorite to dissolve organic debris and disinfect the canal is performed with total volume of 10ml/canal. After the final shaping, the canal is dried with sterile paper points, leaving it ready for medication placement. For the subjects of GI and GII, nano-ketorolac gel and ketorolac gel respectively (Around 2mm3), placed as medicament inside the root canal while those of GIII a placebo gel is placed. Both will be retained for one week. The obturation through cold lateral compaction technique is to be carried out on the next visit.

Randomization and Blinding:

Randomization will be performed using a computer-generated sequence. The patients and outcome assessors will be blinded to the group allocation. Nano-ketorolac production

This study, a formulation containing Ketorolac Tromethamine (KT) at a concentration of 10 mg/mL were developed using Compritol 888 as distinct oleaginous phases. Span 60 was incorporated as a surfactant at a concentration of 1.5%, while the drug-to-oleaginous phase ratio was maintained at 1:2. The Solid Lipid Nanoparticles (SLNs) were formulated using high-shear homogenization to ensure optimal particle size and stability. The nano-Ketorolac will be manufactured in the college of phramaceutical sciences and drug manufacturing, Misr University for Science and Technology, , Egypt.

Statistical Analysis Data will be analyzed using SPSS software. Data will be tested for its normal distribution; accordingly, the appropriate test will be conducted. Statistical significance will be set at p < 0.05.

Ethical Considerations

* The study will be conducted in accordance with the Declaration of Helsinki.
* Ethical approval will be obtained from the Institutional Ethical Committee of Misr University for Science and Technology.
* Informed consent will be obtained from all participants before their inclusion.
* Patients will be informed of their right to withdraw at any time without consequences.
* Data confidentiality will be maintained throughout the study.

Pain management in endodontics has been extensively studied, with a focus on pharmacological interventions, anesthetic techniques, and intracanal medicaments to improve post-operative outcomes. Several studies have explored the effectiveness of NSAIDs, corticosteroids, and advanced anesthetic techniques in controlling pain, but challenges persist, particularly in cases involving necrotic pulp and apical periodontitis.

DETAILED DESCRIPTION:
Study Design: This study will be a randomized, double-blinded, placebo-controlled clinical trial.

Participants and Setting: The study will be conducted at the clinics of Collage of Oral and dental surgery, Misr University for Science and Technology. Patients diagnosed with necrotic pulp and apical periodontitis requiring root canal treatment will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 years.
* Patients who are diagnosed with necrotic pulp and chronic apical periodontitis in a single-rooted tooth.
* Patients who provide written informed consent.
* Patients with no systemic diseases affecting pain perception or wound healing.

Exclusion Criteria:

* Patients with irreversible pulpitis or acute periapical abscess
* Patients with a history of NSAID or opioid use within 24 hours before treatment.
* Pregnant or lactating women.
* Patients who require more than two-visits root canal treatment due to anatomical or pathological factors.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
post-endodontic pain | • Pre-treatment (baseline) • 6 hours post-treatment • 12 hours post-treatment • 24 hours post-treatment • 48 hours post-treatment • 7 days post-treatment
  Pain intensity will be assessed using the Visual Analog Scale (VAS) on a 10-point scale (0 = no pain, 10 = worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Eman Maged Fouad, PHD, Principal Investigator — Lecturer of Endodontics, Collage of Oral and Dental Surgery, Misr University for Science and Technology, Giza, Egypt.
Locations (1):
- Collage of Oral and Dental Surgery, Misr University for Science and Technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar G, Jena S, Manila N, Fareed M, Karobari MI. Incidence of postoperative pain after single-visit and multiple-visit root canal therapy: a systematic review. BMC Oral Health. 2025 Jan 8;25(1):47. doi: 10.1186/s12903-024-05412-1. PMID 39780175